CLINICAL TRIAL: NCT06375265
Title: A Pilot Study of Digital Sleep Optimization for Brain Health Outcomes in Older Surgical Patients (SLEEP-BOOST)
Brief Title: Digital Sleep Optimization for Brain Health Outcomes in Older Surgical Patients
Acronym: SLEEP-BOOST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lei Gao, MBBS, MMSc, Assistant Professor of Anaesthesia, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024P000780-1
Record Dates: First submitted 2024-04-07; First posted 2024-04-19 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Insomnia; Postoperative Delirium; Delayed Neurocognitive Recovery; Postoperative Neurocognitive Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Emergence Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital CBT-I (Experimental): Preoperative digital CBT-I with the CBT-I Coach app for up to 4 weekly sessions and postoperative booster sessions at 2 weeks and 1 month after surgery.
  Interventions: Behavioral: digital Cognitive Behavioral Therapy for Insomnia (dCBT-I)
- Sleep Health Education (Active Comparator): Preoperative sleep health education materials
  Interventions: Behavioral: Sleep Health Education

INTERVENTIONS:
Behavioral: digital Cognitive Behavioral Therapy for Insomnia (dCBT-I) — Preoperative hybrid intervention (in-person or via phone/video) over 4 weeks, and at 2 weeks, and 1 month after surgery using content from the CBT-I Coach app from Veteran Affairs.
  Arms: Digital CBT-I
Behavioral: Sleep Health Education — Sleep Health Education materials provided
  Arms: Sleep Health Education

SUMMARY:
The Sleep Optimization for Brain Health Outcomes in Older Surgical Patients (SLEEP-BOOST) is a pilot randomized, controlled, singled-blinded (participant) trial in major orthopedic joint surgery patients that will build on a previously clinically tested cognitive behavioral therapy for insomnia (CBT-I) mobile application paired with a wearable device (wrist actigraphy).

DETAILED DESCRIPTION:
CBT-I is the frontline treatment for insomnia but is not considered for preoperative care of older surgical patients with insomnia who are at risk of perioperative neurocognitive disorders associated with sleep/circadian dysfunction. We propose to determine if digital CBT-I (dCBT-I) is feasible for treating older surgical patients with insomnia symptoms and to examine the effects of dCBT-I on sleep, cognitive trajectory, mood, pain, activity, and function after surgery. The Sleep Optimization for Brain Health Outcomes in Older Surgical Patients (SLEEP-BOOST) is a pilot randomized, controlled, singled-blinded (participant) trial in major orthopedic joint surgery patients that will build on a previously clinically tested CBT-I mobile application paired with a wearable device (wrist actigraphy).

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 65 years old
2. Scheduled for an elective orthopedic total joint replacement procedure (knee/hip) with an anticipated stay of ≥48 hours
3. At least mild insomnia (ISI score of ≥10 on telephone screening)
4. Stable sleep-affecting medications in the prior month (by clinical review)
5. Own a smart phone
6. Willingness to use the dCBT-I app and actigraphy.

Exclusion Criteria:

1. Current or previous CBT-I
2. Rapidly progressive illnesses/life expectancy <6 months
3. Active psychosis/suicidal ideation
4. Irregular shift work/sleep patterns
5. Moderate-severe sleep apnea (apnea/hypopnea index ≥15) without CPAP compliance per chart review
6. Sleep disorders other than insomnia or apnea
7. Cognitive impairment (diagnosis of dementia)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Adherence | After dCBT-I intervention during Review session ~1 day to 3 weeks before surgery.
  A Patient Adherence Form developed by the Veterans Affairs CBT-I Training Program will be used to assess adherence to the protocol. A mean adherence score across six domains showing good psychometric properties will be derived (0-24; higher represents more adherent)
Insomnia Severity | At screening, baseline, during dCBT-I/control, 2 weeks, 1- and 3-months after surgery
  The Insomnia Severity Index (ISI) questionnaire will be used to determine the quality of sleep for patients (0 to 28; higher represents more severe insomnia symptoms)

SECONDARY OUTCOMES:
Sleep Diary Completion | Throughout the study 3-4 weeks before surgery, and 2 weeks, 1 month and 3 months after surgery.
  The number of days of completed sleep diaries will be recorded.
Homework Completion | After dCBT-I intervention during Review session ~1 day to 3 weeks before surgery.
  The amount of time spent on CBT-I homework will be recorded.
Utility | After dCBT-I intervention during Review session ~1 day to 1 week before surgery.
  A 16-item digital intervention utility questionnaire will be used to assess patient usage of the app (0-64; higher represents more perceived utility)
Satisfaction with intervention | After dCBT-I intervention during Review session ~1 days to 1 week before surgery.
  A 9-item survey will be used to assess which elements of the app were most helpful and the likelihood the patient would recommend it to family/friends.
Cognition | At baseline and 2 weeks, 1- and 3-months after surgery
  Telephonic Montreal Cognitive Assessment (tMoCA) test to assess cognition
Pain severity | At baseline and 2 weeks, 1- and 3-months after surgery
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain will measure functional pain severity
Mood | At baseline and 1- and 3-months after surgery
  The Geriatric Depression Scale-15 will be used to assess the mood of the patients (0-15; higher represents more severe mood/depression symptoms)
Anxiety | At baseline and 1- and 3-months after surgery
  Generalize Anxiety Disorder 7 (GAD-7; 0-21; higher represents more anxiety symptoms)
Function | At baseline and 2 weeks, 1- and 3-months after surgery
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function
Postoperative Delirium Incidence | From postoperative day 1 to postoperative day 3
  The Confusion Assessment Method (3D-CAM) will be used to monitor signs of delirium in patients.
Postoperative Delirium Severity | From postoperative day 1 to postoperative day 3
  The Confusion Assessment Method (CAM)-Severity assessment will be used to monitor signs of delirium severity in patients.
Delayed Neurocognitive Recovery | At 1-months after surgery
  Using cognitive change from baseline (1 standard deviation from the mean).
Postoperative Neurocognitive Disorders (NCD) | At 3-months after surgery
  Using cognitive change from baseline (1 standard deviation from the mean).
Sleep Efficiency | At baseline, immediately after the intervention, and 2 weeks, 1- and 3-months after surgery
  Actigraphy and diary-derived

OTHER OUTCOMES:
Circadian Rest-Activity Rhythms | At baseline, immediately after the intervention, and 2 weeks, 1- and 3-months after surgery
  Motor activity will be recorded on wrist actigraphy watches to derive amplitude, acrophase, interdaily stability, intradaily variability, most active 10h (M10), least active 5h (L5), relative amplitude (RA), fractal motor activity regulation (FMAR).

CONTACTS AND LOCATIONS:
Overall Officials: Lei Gao, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States